CLINICAL TRIAL: NCT02800954
Title: Value of Macrophage-Colony Stimulating Factor as a New Marker of Bone Lesions in Multiple Myeloma
Acronym: MCSF-MYELOME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AOL08-DR-SALLE
Record Dates: First submitted 2016-06-08; First posted 2016-06-15 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; bone lesions; Macrophage-Colony Stimulating Factor
MeSH Terms: conditions — Multiple Myeloma | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- multiple myeloma group (Experimental): case group = patients with multiple myeloma
  Interventions: Biological: blood samples; Biological: Bone marow samples
- MGUS group (Experimental): monoclonal gammopathy of undetermined significance
  Interventions: Biological: blood samples; Biological: Bone marow samples
- healthy control group (Other): control group = healthy subjects
  Interventions: Biological: blood samples

INTERVENTIONS:
Biological: blood samples
Biological: Bone marow samples
  Arms: MGUS group; multiple myeloma group

SUMMARY:
The Primary objective of this study is to compare serum levels of Macrophage-Colony Stimulating Factor (M-CSF) in a population of patients with multiple myeloma (MM), in a population of patients with Monoclonal Gammopathy of Undetermined Significance (MGUS) and in a control population.

ELIGIBILITY:
Inclusion Criteria:

For the multiple myeloma group

* confirmed diagnosis of de novo multiple myeloma according to the International Myeloma Working Group criteria
* bisphosphonate therapy for more than 60 days,
* signature of the informed consent form,
* patients over the age of 18 years. For the monoclonal gammopathy of undetermined significance (MGUS) group
* confirmed diagnosis of MGUS according to the International Myeloma Working Group criteria
* signature of the informed consent form,
* patients over the age of 18 years. For the healthy control group
* signature of the informed consent form,
* subjects over the age of 18 years.

Exclusion Criteria:

* patients with thyroid or parathyroid disease,
* osteomalacia, rheumatoid arthritis, Paget's disease, osteoporosis,
* bisphosphonate therapy for less than 60 days,
* absence of informed consent,
* patients under the age of 18 years.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2009-02-23 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2018-07-10 (Actual)

PRIMARY OUTCOMES:
Serum Macrophage-Colony Stimulating Factor (M-CSF) levels | Day 1

SECONDARY OUTCOMES:
Tumour osteolysis | Day 1
  determined by the presence of osteolytic lesions, osteopenia or pathological fractures, presence of bone pain

CONTACTS AND LOCATIONS:
Overall Officials: Valéry SALLE, PhD, Principal Investigator — CHU Amiens
Locations (3):
- France (3):
  - CHU Amiens, Amiens
  - CH Beauvais, Beauvais
  - Ch Saint Quentin, Saint-Quentin

REFERENCES:
- [Result] From the American Association of Neurological Surgeons (AANS), American Society of Neuroradiology (ASNR), Cardiovascular and Interventional Radiology Society of Europe (CIRSE), Canadian Interventional Radiology Association (CIRA), Congress of Neurological Surgeons (CNS), European Society of Minimally Invasive Neurological Therapy (ESMINT), European Society of Neuroradiology (ESNR), European Stroke Organization (ESO), Society for Cardiovascular Angiography and Interventions (SCAI), Society of Interventional Radiology (SIR), Society of NeuroInterventional Surgery (SNIS), and World Stroke Organization (WSO); Sacks D, Baxter B, Campbell BCV, Carpenter JS, Cognard C, Dippel D, Eesa M, Fischer U, Hausegger K, Hirsch JA, Shazam Hussain M, Jansen O, Jayaraman MV, Khalessi AA, Kluck BW, Lavine S, Meyers PM, Ramee S, Rufenacht DA, Schirmer CM, Vorwerk D. Multisociety Consensus Quality Improvement Revised Consensus Statement for Endovascular Therapy of Acute Ischemic Stroke. Int J Stroke. 2018 Aug;13(6):612-632. doi: 10.1177/1747493018778713. Epub 2018 May 22. No abstract available. PMID 29786478